CLINICAL TRIAL: NCT00352534
Title: Treatment for Very Low and Standard Risk Favorable Histology Wilms Tumor
Brief Title: Vincristine, Dactinomycin, and Doxorubicin With or Without Radiation Therapy or Observation Only in Treating Younger Patients Who Are Undergoing Surgery for Newly Diagnosed Stage I, Stage II, or Stage III Wilms' Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREN0532; NCI-2009-01067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 06-936; AREN0532; CDR0000487540; AREN0532 (Other: Children's Oncology Group); AREN0532 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Stage I Kidney Wilms Tumor; Stage II Kidney Wilms Tumor; Stage III Kidney Wilms Tumor
MeSH Terms: conditions — Wilms Tumor | interventions — Radiotherapy, Conformal; Specimen Handling; X-Rays; Dactinomycin; Doxorubicin; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum I (very low-risk disease) (Experimental): Patients undergo nephrectomy only. If they meet criteria, they are then observed periodically for 5 years. Patients with recurrent disease undergo surgery (immediate or delayed) and receive chemotherapy as in stratum III. Patients with no metachronous renal disease receive radiotherapy. Patients with metachronous disease undergo renal-sparing surgery and chemotherapy as in stratum III, but no radiotherapy. Treatment continues for up to 25 weeks. Additionally, patients undergo chest X-ray, CT or MRI, ultrasound, echocardiography, and blood sample collection throughout the study.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate
- Stratum II (standard-risk, stage I or II) (Experimental): Patients undergo nephrectomy. Between 9 and 14 days post-nephrectomy, patients receive vincristine IV beginning on day 1, every week for 10 weeks then every 3 weeks for a total of 15 doses. Patients receive dactinomycin IV beginning day 1, alternating every 3 weeks with doxorubicin hydrochloride IV for a total of 5 doses of dactinomycin and 4 doses of doxorubicin. Treatment continues for up to 25 weeks. Additionally, patients undergo chest X-ray, CT or MRI, ultrasound, echocardiography, and blood sample collection throughout the study.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate
- Stratum III (standard-risk, stage III) (Experimental): Patients undergo nephrectomy, if feasible, or biopsy. For patients who undergo biopsy only, definitive surgery is undertaken at week 7 or 13. Between 9 and 14 days post-nephrectomy, patients receive vincristine IV beginning on day 1 every week for 10 weeks then every 3 weeks for a total of 15 doses. Patients receive dactinomycin IV beginning day 1, alternating every 3 weeks with doxorubicin hydrochloride IV for a total of 5 doses of dactinomycin and 4 dose of doxorubicin hydrochloride. Patients undergo radiotherapy over 5-7 days after nephrectomy. Treatment continues for up to 25 weeks. Additionally, patients undergo chest X-ray, CT or MRI, ultrasound, echocardiography, and blood sample collection throughout the study.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Patients undergo radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest X-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial is studying vincristine, dactinomycin, and doxorubicin with or without radiation therapy or observation only to see how well they work in treating patients undergoing surgery for newly diagnosed stage I, stage II, or stage III Wilms' tumor. Drugs used in chemotherapy, such as vincristine, dactinomycin, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors.Giving these treatments after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the overall and event-free survival of younger patients with newly diagnosed stage I favorable histology Wilms' tumor (< 2 years of age and < 550gms) treated with nephrectomy only (very low risk), or with newly diagnosed stage III favorable histology Wilms tumor with possible nephrectomy followed by vincristine, dactinomycin, doxorubicin hydrochloride, and radiotherapy (standard risk).

SECONDARY OBJECTIVES:

I. Determine the effects of adding doxorubicin hydrochloride to the regimen for patients with stage I or II favorable histology found to have a high-risk biological marker.

II. Determine whether the omission of adjuvant therapy increases the incidence of contralateral kidney lesions in patients with very low-risk disease treated by nephrectomy and observation only.

III. Determine whether the omission of adjuvant therapy increases the incidence of renal failure in patients with very low-risk disease who have metachronous relapse.

IV. Correlate study outcomes in patients with standard-risk disease with biological data from tissue collections on protocol study COG-AREN03B2.

OUTLINE: This is a multicenter study. Patients are stratified according to clinical and biological risk factors (very low risk vs standard risk).

STRATUM I: (very low-risk disease) Patients undergo nephrectomy only. If they meet criteria, they are then observed periodically for 5 years. Patients with recurrent disease undergo surgery (immediate or delayed) and receive chemotherapy as in stratum III. Patients with no metachronous renal disease receive radiotherapy. Patients with metachronous disease undergo renal-sparing surgery and chemotherapy as in stratum III, but no radiotherapy. Treatment continues for up to 25 weeks.

STRATUM II: (standard-risk, stage I or II disease with adverse biological marker) Patients undergo nephrectomy. Between 9 and 14 days post-nephrectomy, patients receive vincristine IV beginning on day 1, every week for 10 weeks then every 3 weeks for a total of 15 doses. Patients receive dactinomycin IV beginning day 1, alternating every 3 weeks with doxorubicin hydrochloride IV for a total of 5 doses of dactinomycin and 4 doses of doxorubicin. Treatment continues for up to 25 weeks.

STRATUM III: (standard-risk, stage III disease) Patients undergo nephrectomy, if feasible, or biopsy. For patients who undergo biopsy only, definitive surgery is undertaken at week 7 or 13. Between 9 and 14 days post-nephrectomy, patients receive vincristine IV beginning on day 1 every week for 10 weeks then every 3 weeks for a total of 15 doses. Patients receive dactinomycin IV beginning day 1, alternating every 3 weeks with doxorubicin hydrochloride IV for a total of 5 doses of dactinomycin and 4 dose of doxorubicin hydrochloride. Patients undergo radiotherapy over 5-7 days after nephrectomy. Treatment continues for up to 25 weeks.

Additionally, patients undergo chest X-ray, computed tomography (CT) or magnetic resonance imaging (MRI), ultrasound, echocardiography, and blood sample collection throughout the study.

After completion of study treatment, patients are followed periodically for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Wilms' tumor

  * Newly diagnosed stage I-III disease
  * Favorable histology
* No moderate- or high-risk Wilms' predisposition syndromes
* Must meet 1 of the following disease stratification categories:

  * Very low-risk disease

    * Stage I disease
    * Age < 2 years
    * Tumor weight < 550 g
    * Regional lymph nodes histologically negative (must have been sampled)
    * No pulmonary metastases on CT scan of chest
    * No synchronous bilateral Wilms tumors (Stage V)
    * Not predisposed to develop bilateral Wilms tumors, defined as unilateral Wilms tumor and any of the following:

      * Aniridia
      * Beckwith-Wiedemann syndrome
      * Simpson-Golabi-Behmel syndrome
      * Denys-Drash syndrome or other associated genito-urinary anomalies
      * Multicentric WT or unilateral WT with contralateral nephrogenic rest(s) in a child < 1 year of age
      * Diffuse hyperplastic perilobar nephroblastomatosis
  * Standard-risk disease meeting 1 of the following criteria:

    * Disease does not require radiotherapy

      * LOH at chromosomes 1p and 16q for stage I or II
      * Stage I disease meeting 1 of the following criteria:

        * Age ≥ 2 years to age < 30 years
        * Tumor weight ≥ 500 g
      * Stage II disease

        * Age < 30 years
        * Any tumor weight
    * Disease requires radiotherapy

      * No LOH at chromosomes 1p and 16q*
      * Stage III disease
* Must be enrolled on protocol COG-AREN03B2
* Karnofsky performance status (PS) 50-100% for patients > 16 years old
* Lansky PS 50-100% for patients ≤ 16 years old
* Bilirubin (direct) ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram (standard-risk disease)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patient must use effective contraception
* No prior tumor-directed chemotherapy or radiotherapy

  * Patients transferring from AREN03B2 with LOH 1p and 16q allowed

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 808 (Actual)
Dates: Start 2006-11-06 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2025-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mullen, Principal Investigator — Children's Oncology Group
Locations (240):
- United States (210):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (17):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Swiss Pediatric Oncology Group - Bern, Bern, Switzerland

REFERENCES:
- [Derived] Dix DB, Fernandez CV, Chi YY, Mullen EA, Geller JI, Gratias EJ, Khanna G, Kalapurakal JA, Perlman EJ, Seibel NL, Ehrlich PF, Malogolowkin M, Anderson J, Gastier-Foster J, Shamberger RC, Kim Y, Grundy PE, Dome JS; AREN0532 and AREN0533 study committees. Augmentation of Therapy for Combined Loss of Heterozygosity 1p and 16q in Favorable Histology Wilms Tumor: A Children's Oncology Group AREN0532 and AREN0533 Study Report. J Clin Oncol. 2019 Oct 20;37(30):2769-2777. doi: 10.1200/JCO.18.01972. Epub 2019 Aug 26. PMID 31449468
- [Derived] Fernandez CV, Mullen EA, Chi YY, Ehrlich PF, Perlman EJ, Kalapurakal JA, Khanna G, Paulino AC, Hamilton TE, Gow KW, Tochner Z, Hoffer FA, Withycombe JS, Shamberger RC, Kim Y, Geller JI, Anderson JR, Grundy PE, Dome JS. Outcome and Prognostic Factors in Stage III Favorable-Histology Wilms Tumor: A Report From the Children's Oncology Group Study AREN0532. J Clin Oncol. 2018 Jan 20;36(3):254-261. doi: 10.1200/JCO.2017.73.7999. Epub 2017 Dec 6. PMID 29211618
- [Derived] Fernandez CV, Perlman EJ, Mullen EA, Chi YY, Hamilton TE, Gow KW, Ferrer FA, Barnhart DC, Ehrlich PF, Khanna G, Kalapurakal JA, Bocking T, Huff V, Tian J, Geller JI, Grundy PE, Anderson JR, Dome JS, Shamberger RC. Clinical Outcome and Biological Predictors of Relapse After Nephrectomy Only for Very Low-risk Wilms Tumor: A Report From Children's Oncology Group AREN0532. Ann Surg. 2017 Apr;265(4):835-840. doi: 10.1097/SLA.0000000000001716. PMID 27811504

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage I/II: Patients who have either Very Low Risk Disease, Low Risk Stage I or II no LOH, and Standard Risk, Stage I or II with LOH prior to final Risk Group Assignment
- Stage III: Patients who have either Standard Risk, Stage III and High Risk Patients prior to final Risk Group Assignment.
- Very Low Risk Disease: Treatment arm. Nephrectomy and re-evaluation,very low-risk disease.
- Low Risk, Stage I or II, no LOH: Treatment arm. Low risk, stage I or II, no loss of heterozygosity (LOH).
- Standard Risk, Stage I or II With LOH: Treatment arm. Standard Risk, Stage I or II with LOH.
- Standard Risk, Stage III: Treatment arm. Standard Risk, Stage III.
- High Risk: Treatment arm. High risk.
Period: Initial Staging
Arm/Group | Stage I/II | Stage III | Very Low Risk Disease | Low Risk, Stage I or II, no LOH | Standard Risk, Stage I or II With LOH | Standard Risk, Stage III | High Risk
Started | 211 | 597 | 0 | 0 | 0 | 0 | 0
Completed | 203 | 588 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 8 | 9 | 0 | 0 | 0 | 0 | 0
Period: Final Risk Group Assignment
Arm/Group | Stage I/II | Stage III | Very Low Risk Disease | Low Risk, Stage I or II, no LOH | Standard Risk, Stage I or II With LOH | Standard Risk, Stage III | High Risk
Started | 0 | 0 | 119 | 52 | 32 | 548 | 40
Completed | 0 | 0 | 116 | 49 | 31 | 503 | 1
Not Completed | 0 | 0 | 3 | 3 | 1 | 45 | 39
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1 | 19 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 8 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Ineligible | 0 | 0 | 3 | 1 | 0 | 13 | 0
Not completed — Enrollment onto another COG study | 0 | 0 | 0 | 0 | 0 | 0 | 28
Not completed — Stage III Wilms tumor with LOH | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Stage I or II: Patients who have either Very Low Risk Disease, Low Risk Stage I or II no LOH, and Standard Risk, Stage I or II with LOH prior to final Risk Group Assignment. Stage III: Patients who have either Standard Risk, Stage III and High Risk Patients prior to final Risk Group Assignment.
Groups:
- Stage I or II: Patients who have either Very Low Risk Disease, Low Risk Stage I or II no LOH, and Standard Risk, Stage I or II with LOH prior to final Risk Group Assignment.
- Total: Total of all reporting groups
Arm/Group | Stage I or II | Stage III | Total
Number analyzed (Participants) | 211 | 597 | 808
Age, Continuous [Mean (Standard Deviation); unit: Months] | 23.91 (24.37) | 50.62 (30.89) | 43.64 (31.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 318 | 428
  Male | 101 | 279 | 380
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 89 | 127
  Not Hispanic or Latino | 165 | 482 | 647
  Unknown or Not Reported | 8 | 26 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 6 | 7
  Asian | 2 | 15 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 89 | 128
  White | 141 | 417 | 558
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 70 | 98

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Probability
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study.
Time Frame: 4 years
Population: Eligible very low risk or standard risk patients
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- Very Low Risk: Very Low Risk
- Standard Risk, Stage I or II, With LOH: Standard Risk, Stage I or II, with LOH
- Standard Risk, Stage III: Standard Risk, Stage III
Arm/Group | Very Low Risk | Standard Risk, Stage I or II, With LOH | Standard Risk, Stage III
Number analyzed (Participants) | 116 | 32 | 535
Probability | 0.88 [0.79 to 0.98] | 0.87 [0.73 to 1.00] | 0.88 [0.85 to 0.91]

2. Primary Outcome: Overall Survival (OS) Probability
Description: Probability of being alive after 4 years in the study.
Time Frame: 4 years
Population: Eligible very low risk or standard risk patients
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Very Low Risk | Standard Risk, Stage I or II, With LOH | Standard Risk, Stage III
Number analyzed (Participants) | 116 | 32 | 535
Probability | 1.00 [1 to 1] | 1.00 [1 to 1] | 0.97 [0.95 to 0.99]

3. Secondary Outcome: Incidence of Contralateral Kidney Lesions
Description: Number of contralateral kidney lesions during follow-up.
Time Frame: During follow-up
Population: Very low risk patients treated by nephrectomy and observation only.
Measure: Number; unit: Lesions
Arm/Group | Very Low Risk
Number analyzed (Participants) | 116
Lesions | 1

4. Secondary Outcome: Incidence of Renal Failure
Description: Number of renal failures defined as requiring dialysis or renal transplant as determined by low GFR during follow-up
Time Frame: During follow-up
Population: Very low risk patients that have metachronous relapse.
Measure: Number; unit: Incidents
Arm/Group | Very Low Risk
Number analyzed (Participants) | 116
Incidents | 0

ADVERSE EVENTS:
Description: Adverse Events were reported for eligible patients only.
Groups:
- Very Low Risk Disease: Nephrectomy and Re-evaluation
- Low Risk, Stage I or II, no LOH: Low risk, stage I or II, no loss of heterozygosity (LOH).
- Standard Risk, Stage I or II, With LOH: Standard Risk, Stage I or II, with loss of heterozygosity (LOH).
- Standard Risk, Stage III: Nephrectomy/Biopsy, Chemotherapy
- High Risk: High risk.
Arm/Group | Very Low Risk Disease | Low Risk, Stage I or II, no LOH | Standard Risk, Stage I or II, With LOH | Standard Risk, Stage III | High Risk
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/51 | 0/32 | 20/535 | 1/40
Other Adverse Events (participants affected / at risk) | 0/116 | 2/51 | 0/32 | 31/535 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Risk Disease (N=116) | Low Risk, Stage I or II, no LOH (N=51) | Standard Risk, Stage I or II, With LOH (N=32) | Standard Risk, Stage III (N=535) | High Risk (N=40)
24600-Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
37200-General disorders and administration site conditions (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
40000-Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
51900-Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
55700-Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
58000-Neoplasms benign malignant and unspecified (incl cy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
73600-Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
73700-Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Risk Disease (N=116) | Low Risk, Stage I or II, no LOH (N=51) | Standard Risk, Stage I or II, With LOH (N=32) | Standard Risk, Stage III (N=535) | High Risk (N=40)
11600-Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
14900-Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
33900-Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
36400-Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
42500-Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
43600-Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
44800-Infections and infestations - Other specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
47000-Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
58300-Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 7 (9) | 0 (0)
66800-Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
71300-Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
71600-Respiratory thoracic and mediastinal disorders - Ot (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
73700-Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
79600-Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
87900-Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other